CLINICAL TRIAL: NCT01181713
Title: Antibiotic Resistance of Ocular Surface Flora After Continued Use of Topical Antibiotics Post Intravitreal Injections
Brief Title: Change in Ocular Flora Resistance From Repeated Topical Antibiotic Use
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Dr. Peter Kertes, chief, department of ophthalmology, Sunnybrook Health Sciences Centre
Other Study IDs: SBK-OcuFResis
Record Dates: First submitted 2010-02-08; First posted 2010-08-13 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Increased Drug Resistance; Infection Resistant to Quinolones and Fluoroquinolones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No Antibiotic: No prophylactic antibiotic post intravitreal injection
- Prophylactic Antibiotic: Group treated with 3 day course of prophylactic topic antibiotic, fourth generation fluoroquinolones, after each intravitreal injection

SUMMARY:
The purpose of this study is to determine if antibiotic resistance of the ocular surface flora to the 4th generation fluoroquinolones will increase after repeated use of topical antibiotics for three days post intravitreal injection.

DETAILED DESCRIPTION:
Treatment with intravitreal (IVT) injections has increased during the last several years as evidence has accumulated demonstrating the efficacy of anti-vascular endothelial growth factor agents in the treatment of neovascular age-related macular degeneration (AMD) and various retinal vascular diseases.

Although IVT injections are generally safe, infectious endophthalmitis is a rare but devastating complication, and the risk of morbidity and vision loss from endophthalmitis is high. The objective is to examine the change in antibiotic resistance of ocular surface flora with repeated prophylactic use of antibiotics after IVT injection for AMD.

Yin, V. T., Weisbrod, D. J., Eng, K. T., Schwartz, C., Kohly, R., Mandelcorn, E., Lam, W., Daneman, N., Simor, A., & Kertes, P. J. (2013). Antibiotic resistance of ocular surface flora with repeated use of a topical antibiotic after intravitreal injection. JAMA ophthalmology, 131(4), 456-461.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for intravitreal injection for neovascular age-related macular degeneration (ARMD)
* 65 years or older
* able to provide informed consent.

Exclusion Criteria:

* diagnosed with an active ocular, periocular or systemic infection
* previously received treatment with an intravitreal injection
* previously treated with antibiotics in the past three months
* unable to attend the scheduled follow-up appointments or to complete treatment for any reason

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient recruitment would be from the Sunnybrook Health and Sciences Centre Department of Ophthalmology
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
ocular flora resistance to 4th generation fluoroquinolone | 1 year
  Outcome will examine the change in amount, type and antibiotic resistance profile of ocular surface flora over the 3 months. Charcoal swab of the conjunctiva will be cultured, organisms grown will be identified and resistance to moxifloxacin will be quantified by minimal inhibitory resistance (MIC).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kertes, MD, FRCSC, Study Chair — Sunnybrook Health Sciences Centre; Vivian T Yin, MD, Study Director — University of Toronto; Daniel Weisbrod, MD, FRCSC, Study Director — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health and Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Yin VT, Weisbrod DJ, Eng KT, Schwartz C, Kohly R, Mandelcorn E, Lam WC, Daneman N, Simor A, Kertes PJ. Antibiotic resistance of ocular surface flora with repeated use of a topical antibiotic after intravitreal injection. JAMA Ophthalmol. 2013 Apr;131(4):456-61. doi: 10.1001/jamaophthalmol.2013.2379. PMID 23430175